CLINICAL TRIAL: NCT06044090
Title: Neuroinflammatory Mechanisms Linking Chronic Stress to Motivational Deficits
Brief Title: Brain and Stress Study
Acronym: BASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-3111
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-04

CONDITIONS: Stress, Psychological; Motivation
MeSH Terms: conditions — Stress, Psychological | interventions — Minocycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo followed by Minocycline (Experimental): In this arm, participants will take a 5-day course of placebo-control pills and then a 5-day course of 200 mg of minocycline. Sessions will be separated by a minimum washout period of 14 days.
  Interventions: Drug: Minocycline; Drug: Placebo
- Minocycline followed by Placebo (Experimental): In this arm, participants will take a 5-day course of 200 mg of minocycline and then a 5-day course of placebo-control pills. Sessions will be separated by a minimum washout period of 14 days.
  Interventions: Drug: Minocycline; Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Participants will take 2 pills of 100 mg totaling a 200 mg dose of minocycline per day.
  Other Names: Minocin, Solodyn, Ximino, CoreMino
Drug: Placebo — A placebo is a sugar pill that has no therapeutic effect and will be administered orally. Participants will receive 2 placebo tablets matching the Minocycline tablets daily for 5 days.
  Other Names: sugar pill

SUMMARY:
Motivational deficits such as anhedonia are core to several psychiatric disorders and underlie significant functional impairment. This double-blind, placebo-controlled crossover trial of minocycline, an anti-[neuro]inflammatory agent, examines links between chronic stress and responses to a reward-related motivation task. It will evaluate the effects of pharmacologically attenuating neuroinflammation on behavioral responses to a reward-related motivation task in individuals experiencing unemployment. Understanding the effects of neuroinflammation on reward function among individuals experiencing chronic stress represents a critical first step in identifying novel neuroimmune targets for future clinical trials.

DETAILED DESCRIPTION:
This study seeks to conduct translational work that extends rich preclinical findings to the clinical domain to validate whether neuroinflammatory dysregulation is strongly tied to anhedonia. This project addresses critical gaps in the scientific literature by recruiting a chronically stressed sample of individuals-employment seeking individuals who report significant stress-- and will use an experimental therapeutics approach to attenuate neuroinflammation and assess behavioral changes in motivation.

One major obstacle in understanding how neuroinflammation influences motivation involves technological challenges such that conventional approaches are invasive, expensive, and/or lacking specificity. Although static levels of neuroinflammation in humans have been measured via cross sectional studies, capturing behavioral shifts following experimental manipulation has not been done. This gap limits the ability to develop a more precise understanding of how neuroinflammation causes motivational deficits in humans. The proposed project will employ a mechanistic clinical trial of the anti-[neuro]inflammatory agent, minocycline, to address these limitations. In animal models, minocycline has attenuated the deleterious effects of neuroinflammation on neurogenesis, long-term potentiation, and neuronal survival. This study will extend research to humans to examine whether links between neuroinflammation and behavioral responses to a reward-related motivation task differ among chronically stressed individuals taking minocycline and the placebo control. The proposed project will provide preliminary evidence for potential neural targets that have relevance for motivational deficits due to neuroinflammation.

Once screening is complete, participants will come to UNC to complete quality-of-life surveys, learn about the full study schedule, and receive the first dose of medication. This visit will last about 90 minutes. Participants will be asked to participate in two medication periods, meaning they will take both minocycline (antibiotic medication) for 5-days, and an inactive substance (placebo sugar pill) for 5-days. This will investigate whether there are changes in their responses to negative and positive information. After taking the first medication for five days, participants will come in to complete a computer task (Probabilistic Reward Task) and some follow-up surveys (Snaith-Hamilton Pleasure Scale and Motivation and Pleasure Scale). This visit will last about 90 minutes. Participants will then get at least a 2-week break before taking the second medication for five days. Then, they will come back for another 90-minute visit to complete the same computer task and follow-up surveys. The total study duration including the break is about one month. The total time in study sessions on campus over the month will be 4.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* 25-60 years old
* Unemployed (working less than 20 hours per week)
* Have been unemployed for at least 6 months
* Seeking employment
* Having trouble finding a job (i.e., actively seeking and applying for jobs but not successful in landing a job)
* Reports greater than 5 points on Job Stress Items
* Regular access to a mobile phone

Exclusion Criteria:

* Self-reported physical illnesses: diabetes, cardiovascular diseases, high blood pressure, inflammatory bowel diseases, rheumatoid arthritis, asthma, autoimmune disease, Crohn's disease, ulcerative colitis, lupus
* neurological conditions (e.g., Traumatic Brain Injury, stroke)
* pregnant (as measured by urine pregnancy screen) or breastfeeding
* current use of psychotropic medications
* Current regular recreational drug or alcohol use (i.e., 4 or more times per week)
* chronic diseases that significantly impact inflammatory markers (e.g., cancer)
* known allergies or hypersensitivities to tetracycline antibiotics, aspirin or other NSAIDs
* current antibiotic use
* regular use of steroidal or non-steroidal anti-inflammatory medications (i.e., 2 or more times a week)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Alvarez, PhD, Study Director — University of North Carolina, Chapel Hill; Keely Muscatell, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Howell Hall, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Kangas BD, Der-Avakian A, Pizzagalli DA. Probabilistic Reinforcement Learning and Anhedonia. Curr Top Behav Neurosci. 2022;58:355-377. doi: 10.1007/7854_2022_349. PMID 35435644
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Llerena K, Park SG, McCarthy JM, Couture SM, Bennett ME, Blanchard JJ. The Motivation and Pleasure Scale-Self-Report (MAP-SR): reliability and validity of a self-report measure of negative symptoms. Compr Psychiatry. 2013 Jul;54(5):568-74. doi: 10.1016/j.comppsych.2012.12.001. Epub 2013 Jan 22. PMID 23351831

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (5 Days)
Arm/Group | Placebo Followed by Minocycline | Minocycline Followed by Placebo
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Placebo Followed by Minocycline | Minocycline Followed by Placebo
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Second Intervention (5 Days)
Arm/Group | Placebo Followed by Minocycline | Minocycline Followed by Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Individuals who completed at least one treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Response Bias During the Probabilistic Reward Task
Description: The aim of Probabilistic Reward Task (PRT) is to win as much money as possible by correctly identifying the presence of a short versus long mouth on a cartoon face. The task aims to produce a response bias toward the mouth length that is more often positively reinforced. The response bias score is a ratio of the number of times the participant chooses the high reward versus the low reward stimulus. Scores range from -1 to +1, with a positive score indicating a stronger bias toward the high reward stimulus.
  The change in response bias is calculated by subtracting response bias during the PRT in the placebo condition from the minocycline condition. This difference measures an individual's change in reward behavior after a 5-day dosage of an anti-neuroinflammatory agent.
Time Frame: within approximately 24 hours after the final dose; Day 6 minocycline to Day 6 placebo
Measure: Mean (Standard Deviation); unit: Ratio (Response Bias Score)
Groups:
- Minocycline: In this arm, participants will take a 5-day course of 200 mg of minocycline.
  Minocycline: Participants will take 2 pills of 100 mg totaling a 200 mg dose of minocycline per day.
- Placebo: In this arm, participants will take a 5-day course of placebo-control pills.
  Placebo: A placebo is a sugar pill that has no therapeutic effect and will be administered orally. Participants will receive 2 placebo tablets matching the Minocycline tablets daily for 5 days.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 8
Ratio (Response Bias Score) | 0.195 (0.206) | 0.203 (0.199)
Statistical Analysis 1: Comparison: Minocycline; Test type: Superiority; p = 0.856, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.613, t-test, 2 sided

2. Secondary Outcome: Change in Snaith Hamilton Pleasure Scale Score
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) is a tool to assess symptoms of reduced motivation. The SHAPS uses 14 questions, each rated on a Likert scale of 1-4. The total score on the scale ranges from 14-56, with lower scores reflecting lower motivation. Scores will be compared across conditions to determine whether motivation changes in the minocycline condition as compared to the placebo.
Time Frame: within approximately 24 hours after the final dose; Day 6 minocycline to Day 6 placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 8
score on a scale | 3.286 (1.590) | 2.933 (1.580)
Statistical Analysis 1: Comparison: Minocycline; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.691, t-test, 2 sided

3. Secondary Outcome: Change in Motivation and Pleasure Scale (MAPS) Score
Description: The Motivation and Pleasure Scale (MAP) will be used to capture self-reported aspects of reduced motivation. The scale uses 18 questions, each rated on a Likert scale of 0-4. The total score on the scale ranges from 0-72, with lower scores reflecting lower motivation. Scores will be compared across conditions to determine whether motivation changes in the minocycline condition as compared to the placebo.
Time Frame: within approximately 24 hours after the final dose; Day 6 minocycline to Day 6 placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 10 | 8
score on a scale | 37.786 (10.984) | 39.267 (12.870)
Statistical Analysis 1: Comparison: Minocycline; Test type: Superiority; p = 0.225, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.667, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Primary systematic adverse event collection occurred during the two 5-day treatment periods. Any non-systematic adverse event occuring during washout was included. The overall collection period was a combined total of 24 days.
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 8/10 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=10) | Placebo (N=8)
Nausea (Gastrointestinal disorders) | 3 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (7) | 0 (0)
Loss of Appetite (Gastrointestinal disorders) | 5 (6) | 1 (1)
Stomach Ache (Gastrointestinal disorders) | 0 (0) | 1 (4)
Stomach Pain (Gastrointestinal disorders) | 2 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (4) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 0 (0)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Interrupted Sleep (General disorders) | 1 (1) | 0 (0)
Night Terrors (General disorders) | 1 (1) | 0 (0)
A sense of unrealness (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
General Discomfort (General disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT06044090/Prot_SAP_000.pdf